CLINICAL TRIAL: NCT00744536
Title: Revlimid®, and Metronomic Melphalan in the Management of Higher Risk Myelodysplastic Syndromes (MDS) and CMML: A Phase 2 Study"
Brief Title: Efficacy Study of Revlimid® and Low Dose Continuously Administered Melphalan to Treat High Risk MDS
Acronym: REMMYDYS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Celgene (Industry)
Responsible Party: Principal Investigator, Dr. Rena Buckstein, Head Hematology Site Group, Sunnybrook Health Sciences Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RV-MDS-PI-128
Record Dates: First submitted 2008-08-29; First posted 2008-09-01 (Estimated); Last update posted 2017-06-09 (Actual); Status verified 2017-06

CONDITIONS: Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic; Angiogenesis
Keywords: Myelodysplastic syndrome; Chronic myelomonocytic leukemia; High intermediate risk and high risk IPSS score; Angiogenesis; Metronomic chemotherapy; Myelodysplastic Myeloproliferative Diseases
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic; Myelodysplastic-Myeloproliferative Diseases | interventions — Lenalidomide; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Lenalidomide and Melphalan (Experimental): Lenalidomide + Melphalan both given metronomically
  Interventions: Drug: Lenalidomide and melphalan

INTERVENTIONS:
Drug: Lenalidomide and melphalan — Lenalidomide (Revlimid) 10 mg po daily for 21d/28 Melphalan (Melphalan) 2 mg po daily for 21d/28
  Other Names: Revlimid; Melphalan

SUMMARY:
Angiogenesis increases in higher risk MDS patients and those with proliferative CMML. Angiogenesis is associated with increased risk of leukemic transformation and poorer prognoses. Low dose chemotherapy may have anti-angiogenic properties by targetting the genetically stable endothelial cells. Lenalidomide has been recently shown to be highly effective as monotherapy in low/low-intermediate risk MDS, particularly in the subgroup harboring a 5q- deletion. Lenalidomide has not been well studied in higher risk MDS although there are some reports of lenalidomide's efficacy in RAEB-T and AML. One potential mode of action of lenalidomide is inhibition of angiogenesis. The investigators hypothesize that by combining lenalidomide with low dose melphalan in higher risk MDS the investigators will more effectively block angiogenesis and achieve responses or hematologic improvement in MDS.

DETAILED DESCRIPTION:
STUDY OBJECTIVES:

Primary:

1. Determine the overall response rates of low dose melphalan used in combination with lenalidomide in higher risk MDS

Secondary:

1. Determine the frequency of hematologic improvement of low dose melphalan used in combination with lenalidomide in higher risk MDS·
2. Determine the safety and tolerability of low dose melphalan used in combination with lenalidomide in higher risk MDS·
3. Determine the effects of low dose melphalan used in combination with lenalidomide on biomarkers of angiogenesis in higher risk MDS·
4. Determine the frequency of cytogenetic remissions of low dose melphalan used in combination with lenalidomide in higher risk MDS

STUDY DESIGN:

This study is a single center, open-label, non-randomized Phase II study. Patients with higher risk MDS are included. This patient population will be defined by either high intermediate or high risk IPSS scores or proliferative CMML with symptomatic cytopenias or hypersplenism (IPSS score does not apply). If cytogenetics are unavailable, patients with transfusion dependent RAEB-1 will be eligible.

This is an open label, single center non-randomized Phase II study of melphalan 2 mg po and lenalidomide, 10 mg po daily on days 1 - 21 of a 28 day cycle in adult patients with higher risk MDS. Patients may continue to receive drug for a maximum of 12 months or until one of the following occur: death; disease progression (for definition, see appendix D); intercurrent illness that prevents further administration of treatment; unacceptable adverse event(s); patient decides to withdraw from the study; or if general or specific changes in the patient's condition make the patient unsuitable for further treatment, or if after 4 cycles the patient is not deriving clinical benefit from the treatment in the judgment of the investigator. After 12 months, responding patients may continue on oral lenalidomide alone daily (at the dose tolerated by the patient) for 21 days of a 28 day cycle until disease progression, toxicity or death.

Response to treatment and disease progression will be assessed by collecting and evaluating bone marrow aspirates within 10 days of the first dose of cycles 3 and 5 and every three cycles thereafter (every 12 weeks) until confirmation of a complete response. Once confirmed 1 month later, patients will not undergo bone marrow assessments until there is evidence of progression.

Blood tests will include weekly CBC with differential and platelet count, electrolytes, BUN and creatinine for the first 8 weeks, then every 2 weeks until on stable doses, then every 4 weeks thereafter or as clinically indicated. Liver profile will be measured monthly. Bone marrow biopsies/aspirates will be centrally reviewed during or at the end of the study. Approximately 30 days after receiving the last dose of study drug, patients will be reassessed for toxicity, patient status and relapse/progression if applicable. Thereafter, patients will be re-assessed every 3 months until death or loss to follow-up.

Biomarkers of angiogenesis will be measured at the following frequencies: CECs and CEPs at baseline, monthly x 3 then q 3 monthly x 2 then at time of progression or coming off study.Marrow and peripheral blood soluble VEGF and VEGFR-1 and 2 will be measured by ELISA at the same frequency as the bone marrows.Cytogenetics will be performed at baseline, at 3 months and at completion of the study.

STUDY DURATION: 12 months for lenalidomide + melphalan; option to remain on lenalidomide alone if ongoing response at 12 months TOTAL SAMPLE SIZE: 20

ELIGIBILITY:
Inclusion Criteria:

1. Understand and voluntarily sign an informed consent form.
2. Age 18 years or older at the time of signing the informed consent form.
3. Able to adhere to the study visit schedule and other protocol requirements.
4. Must have a diagnosis of high-intermediate or high risk MDS (de novo or secondary) or CMML fitting any of the following classifications (including CMML with wbc < 12,000 x 109/L) and IPSS > 1.5 or proliferative form of CMML (wbc > 12,000 x 109/L for which the IPSS does not apply). If the patient has unsuccessful cytogenetics, patients with WHO classification of transfusion dependent RAEB-1 will be eligible (see appendix B and C for WHO MDS classification).
5. All previous cancer therapy, including radiation, hormonal therapy and surgery, must have been discontinued at least 4 weeks (6 weeks for 5-Azacitidine or bone marrow transplant) prior to treatment in this study.
6. ECOG performance status of <= 2 at study entry (see Appendix A).
7. Laboratory test results within these ranges:

   * Serum calcium <3.0 mmol/L
   * Serum creatinine < 1.5 mg/dL
   * Total bilirubin < 1.5 mg/dL
   * AST (SGOT) and ALT (SGPT) < 2 x ULN

Exclusion Criteria:

1. Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
2. Pregnant or breast-feeding females. (Lactating females must agree not to breast feed while taking lenalidomide).
3. Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
4. Use of any other experimental drug or therapy within 28 days of baseline.
5. Known hypersensitivity to thalidomide or melphalan.
6. The development of erythema nodosum is characterized by a desquamating rash while taking thalidomide or similar drugs.
7. Any prior use of lenalidomide.
8. Concurrent use of other anti-cancer agents or treatments.
9. Known positive for HIV or infectious hepatitis, types A, B or C.
10. Must not have a diagnosis of AML (> 20% blasts) or other progressive malignant disease
11. Must not have received treatment with, erythropoietin, or granulocyte colony-stimulating factors within seven days of study initiation (21 days for pegfilgrastim or Aranesp). Note: use of corticosteroids (topical and inhaled) is permitted and prophylactic steroids are allowed for transfusion reactions, but ongoing oral corticosteroids are not permitted.
12. Serious or non-healing wound, ulcer, or bone fracture.
13. History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 28 days of treatment.
14. Any history of cerebrovascular accident (CVA) or transient ischemic attack within 12 months prior to study entry.
15. Histories of myocardial infarction, cardiac arrhythmia, stable/unstable angina, symptomatic congestive heart failure, or coronary/peripheral artery bypass graft or stenting within 12 months prior to study entry.
16. History of pulmonary embolism within the past 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-01; Primary Completion 2012-01 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate (RR) (as defined by modified international working group standardized response criteria) | 3 years
  Overall Response Rate (RR) (as defined by modified international working group standardized response criteria).

SECONDARY OUTCOMES:
Percent with hematologic improvement | 3 years
  Percent with hematologic improvement.
Percent with cytogenetic remission | 3 years
  Percent with cytogenetic remission.
Overall, progression-free and leukemia-free-survival | 3 yrs
  Overall, progression-free and leukemia-free-survival.
Percent reduction in baseline biomarkers of angiogenesis including: circulating endothelial cells (CEC) and precursors (CEP), plasma and marrow VEGF and VEGFR 1-2 levels | 3 yrs
  Percent reduction in baseline biomarkers of angiogenesis including: circulating endothelial cells (CEC) and precursors (CEP), plasma and marrow VEGF and VEGFR 1-2 levels.
Safety (type, frequency, severity, and relationship of adverse events to study therapy) | 3 yrs
  Safety (type, frequency, severity, and relationship of adverse events to study therapy).

CONTACTS AND LOCATIONS:
Overall Officials: Rena J Buckstein, MD FRCPC, Principal Investigator — Odette Cancer Center
Locations (1):
- Sunnybrook Health Sciences Centre, Odette Cancer Center, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Buckstein R, Kerbel R, Cheung M, Shaked Y, Chodirker L, Lee CR, Lenis M, Davidson C, Cussen MA, Reis M, Chesney A, Zhang L, Mamedov A, Wells RA. Lenalidomide and metronomic melphalan for CMML and higher risk MDS: a phase 2 clinical study with biomarkers of angiogenesis. Leuk Res. 2014 Jul;38(7):756-63. doi: 10.1016/j.leukres.2014.03.022. Epub 2014 Apr 5. PMID 24819395
- See also: Published online to Leukemia Research — http://dx.doi.org/10.1016/j.leukres.2014.03.022